CLINICAL TRIAL: NCT06203171
Title: Preoperative Evaluation: Impact on Perioperative Complications
Brief Title: Preoperative Evaluation on Perioperative Complications
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SUKAEK-2023 17/16
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Complication
Keywords: Anesthesia; preoperative assesment; Perioperative complications
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group C: Patients with perioperative complications
  Interventions: Other: Observational
- Group non-C: Patients with no perioperative complications
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Routine laboratory parameters requested from patients; Direct lung Radiograph and Electrocardiography results were evaluated and preoperative consultations and recommendations requested from the patients were recorded. Type of anesthesia, operation performed, operation duration, intraoperative blood and fluid losses, intraoperative and postoperative complications that develop within the first 24 hours, additional problems that develop (pain, postoperative nausea and vomiting, hypothermia, change of consciousness, bleeding and unplanned transfer to the intensive care unit). postanesthesia recovery The length of stay in the room, length of hospital stay, and method of discharge were recorded. The effects of preoperative laboratory, imaging methods and required consultations on intraoperative and postoperative complications in the first 24 hours were evaluated.

SUMMARY:
Failure to properly manage the perioperative period of patients is associated with increased morbidity and mortality. Preoperative evaluation in patients planned for surgery contributes to reviewing possible perioperative risks, optimizing the patient's functional and physiological status, and reducing the possibility of perioperative complications. Assessments made during the preoperative evaluation process can be used to educate the patient, organize resources for perioperative care, and formulate plans for intraoperative care, postoperative recovery, and perioperative pain management. However, the effect of preoperative evaluation on patient outcomes has not been clearly demonstrated. In this study, the effect of preoperative anesthesia evaluation on perioperative complications was investigated.

DETAILED DESCRIPTION:
Not managing patients well before, during, and after surgery can lead to more health problems and deaths. In wealthy countries, 3-16% of patients face major issues during this time, and 0.4-0.8% of them might end up permanently disabled or dead. Checking patients before surgery helps identify risks, improves their health and fitness, and lowers the chances of problems during this period.

On another note, even though the right surgeries can save lives and prevent injuries, the growing cost of healthcare is a big issue worldwide. In the United States, the rising cost is a concern for everyone, including insurance companies and drug makers. It's believed that treatments that don't really help could be causing about 30% of these high costs.

No matter the surgery, patient's health, or anesthesia plan, checking patients before surgery is key to safe anesthesia for people of all ages. A thorough check before surgery helps manage patient care during this period, prevents surgery cancellations due to patient issues, and helps keep the surgery schedule efficient and cost-effective.

There's no agreed-upon definition for checking patients before anesthesia in medical literature. This check involves looking at the patient's medical history, interviews, physical exams, and test results. Anesthesiologists might also talk to other healthcare workers for more information or help with anesthesia care during this period. The information gathered can help educate the patient, plan for care during and after surgery, and manage pain.

However, it's not clear how much these pre-surgery checks actually improve patient outcomes. A recent study found that seeing a doctor before surgery didn't reduce, but actually increased, the chances of problems after surgery. This study looks at how well pre-surgery anesthesia checks at our center help prevent problems during this period

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* ASA ≤ 3 patients
* Patients over 18 years of age

Exclusion Criteria:

* Emergency surgeries
* ASA > 3 patients
* Pregnant women
* Age > 80
* Age < 18

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo elective surgery have been evaluated by an anesthesiologist at the anesthesia clinic before surgery and have completed the examinations and necessary consultations requested by the anesthesiologist.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Perioperative hemodynamic complications | Up to 24 hours
  New developments in the perioperative period hemodynamic complications
  1. Hypertension; systolic arterial pressure >160 mm Hg
  2. Hypotension; mean arterial pressure < 65 mmHg
  3. Cardiac arrhythmia
  4. Acute Coronary syndrome; ECG changes and/or cardiac enzyme elevation accompanied by chest pain
New developments in the perioperative period respiratuary complications | Up to 24 hours
  Respiratory Failure; Oxygen saturation < 90 or tachypnea (respiratory rate > 20/min

SECONDARY OUTCOMES:
Time of hospital | 2 weeks
  Time in hospital after surgery

CONTACTS AND LOCATIONS:
Overall Officials: OZGUR KOMURCU, 1, Principal Investigator — Samsun University
Locations (1):
- Samsun University, Samsun, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Rose J, Weiser TG, Hider P, Wilson L, Gruen RL, Bickler SW. Estimated need for surgery worldwide based on prevalence of diseases: a modelling strategy for the WHO Global Health Estimate. Lancet Glob Health. 2015 Apr 27;3 Suppl 2(Suppl 2):S13-20. doi: 10.1016/S2214-109X(15)70087-2. PMID 25926315
- [Background] Siddaiah H, Patil S, Shelvan A, Ehrhardt KP, Stark CW, Ulicny K, Ridgell S, Howe A, Cornett EM, Urman RD, Kaye AD. Preoperative laboratory testing: Implications of "Choosing Wisely" guidelines. Best Pract Res Clin Anaesthesiol. 2020 Jun;34(2):303-314. doi: 10.1016/j.bpa.2020.04.006. Epub 2020 Apr 22. PMID 32711836
- [Background] Colla CH, Morden NE, Sequist TD, Schpero WL, Rosenthal MB. Choosing wisely: prevalence and correlates of low-value health care services in the United States. J Gen Intern Med. 2015 Feb;30(2):221-8. doi: 10.1007/s11606-014-3070-z. Epub 2014 Nov 6. PMID 25373832
- [Background] Beckerleg W, Kobewka D, Wijeysundera DN, Sood MM, McIsaac DI. Association of Preoperative Medical Consultation With Reduction in Adverse Postoperative Outcomes and Use of Processes of Care Among Residents of Ontario, Canada. JAMA Intern Med. 2023 May 1;183(5):470-478. doi: 10.1001/jamainternmed.2023.0325. PMID 36972037
- [Derived] Komurcu O, Genc C, Kurt BC, Demir O, Akbas A, Akyurt D, Kusderci HS, Tulgar S, Suren M. Preoperative evaluation: Impact on early perioperative hemodynamic and respiratory complications. BMC Anesthesiol. 2024 Nov 27;24(1):435. doi: 10.1186/s12871-024-02821-1. PMID 39604844